CLINICAL TRIAL: NCT04882410
Title: Extracorporeal CO2 Removal in Acute Exacerbation of COPD Not Responding to Non-Invasive Ventilation: a Single Center Experience
Brief Title: Extracorporeal CO2 Removal in Acute Exacerbation of COPD Not Responding to Non-Invasive Ventilation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Principal Investigator, SILVA, Principal Investigator, Centre Hospitalier de Saint-Denis
Other Study IDs: 0004_CohorteECCO2R
Record Dates: First submitted 2021-04-02; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: COPD Exacerbation Acute
Keywords: Extracorporeal carbon-dioxide removal; ECCO2R; Acute Exacerbation; Chronic Obstructive Pulmonary Disease; Mechanical Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Acute exacerbation of chronic obstructive pulmonary disease (ae-COPD) has a gold standard treatment: non-invasive ventilation (NIV). However, this treatment sometime fails, and an invasive mechanical ventilation (IMV) is required. The extracorporeal CO₂ removal (ECCO₂R) device can be an alternative to intubation. The aim of the study is to evaluate ECCO₂R efficiency and safety and enlighten ECCO₂R benefit/risk compared to IMV.

Methods: Successive ae-COPD patients for whom NIV failed were retrospectively analyzed during two periods: before and after the ECCO₂R device implementation in our ICU in 2015. We considered the before period as standard of care and patients were treated with IMV. The ECCO₂R device was a pump-driven veno-venous system (Xenios AG).

DETAILED DESCRIPTION:
The study compare 2 strategies for COPD patients not responding to non invasive ventilation: the gold standard which is mechanical ventilation and a new technique which is extracorporeal CO2 removal. This technique have been implemented in februrary 2015 in our intensive care unit so we choose to compare patients' outcome before and after the arriving of this device.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* no improvement or worsening of respiratory acidosis after more than one hour of non invasive ventilation treatment
* and non improvement of respiratory distress signs
* and pH < 7,35 and PaCO2 > 45 mmHg

Exclusion Criteria:

* patients not eligible for endotracheal intubation because of ethical limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Successive ae-COPD patients for whom non-invasive ventilation failed during two periods: before and after the ECCO2R device implementation in our ICU in 2015.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Need for invasive mechanical ventilation despite ECCO2R technique | From the begining of the ECCO2R treatment until the end of the ICU hospitalization, up to 6months
  Rate of patients who needed invasive mechanical ventilation despite ECCO2R technique

SECONDARY OUTCOMES:
ECCO2R efficiency | During the treatment up to 6months
  pH
ECCO2R efficiency | During the treatment up to 6months
  PaCO2
Adverse Effects related to ECCO2R and invasive mechanical ventilation during the ICU hospitalization | During the ICU hospitalization up to 6months
  Rate of complications related to ECCO2R and invasive mechanical ventilation: hemorrhagic, thrombotic, haemodynamic, ventilator associated pneumonia, self extubation, death
ICU and hospital length of stay | From the entrance in ICU until the end of hospitalization in ICU and hospital up to 6months
  Length of stay in ICU and hospital
Mortality at day 28 and day 90 | From the entrance in ICU until day 90
  Mortality at day 28 and day 90

REFERENCES:
- [Derived] Azzi M, Aboab J, Alviset S, Ushmorova D, Ferreira L, Ioos V, Memain N, Issoufaly T, Lermuzeaux M, Laine L, Serbouti R, Silva D. Extracorporeal CO2 removal in acute exacerbation of COPD unresponsive to non-invasive ventilation. BMJ Open Respir Res. 2021 Dec;8(1):e001089. doi: 10.1136/bmjresp-2021-001089. PMID 34893522